CLINICAL TRIAL: NCT01231490
Title: A Double Blind, Randomised, Placebo Controlled Methodological Cross-over Study to Investigate the Senstivity of a Novel Study Design and Endpoints to Treatment Effects of Naproxen in Osteoarthritis
Brief Title: Acute Osteoarthritis Experimental Model Study.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: E.D. Derilus; Clinical Disclosure Advisor, GSK Clinical Disclosure
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 111293
Record Dates: First submitted 2010-10-28; First posted 2010-11-01 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: Naproxen
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Naproxen — Capsule
  Arms: Active

SUMMARY:
This is a methodological study designed to investigate a new model for testing pain agents in the treatment of patients with osteoarthritis (OA). This will be a double-blind, randomised, placebo controlled three-way cross-over study in patients with OA of the knee.

DETAILED DESCRIPTION:
The study will include an interim analysis after approximately 50 patients have been randomised. Up to 100 patients with painful Osteoarthritis (OA) of the knee may be recruited into the study. Eligible subjects will wash out of all treatments for their OA pain for a minimum of 7 days apart from protocol rescue medication (paracetamol). Following this, subjects will participate in three short term treatment periods with repeated administration of Naproxen (500 mg/twice daily) or placebo for 3 days. Between treatment periods subjects will receive placebo. Endpoints will include objective assessments of function (time to walk and stair climbing) and subjective assessments of pain including current pain, the Western Ontario and McMaster Universities Arthritis Index (WOMAC) and Patient Global Impression of Change. Throughout the study subjects will be asked to rate their pain periodically. Subjects will attend the unit on Day 1 to be dispensed with study medication and to take their first dose in the unit. They will then return to the unit on Days 8, 10, 15, 17, 22 and 24 for pain assessments, with medication dispensed at each of these visits, excluding Day 24.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of OA of the knee and suitable for the study as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
2. Male or female between 50 to 75 years of age inclusive.
3. A female subject is eligible to participate if she is of non-childbearing potential defined as:

   * Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory].
   * Females with menopausal status ( > 12 months of spontaneous amenorrhea) and receiving hormone replacement therapy (HRT) treatment for more than 3 months.
4. BMI within the range 15-35 kg/m2 (inclusive).
5. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
6. QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.
7. Diagnosis

   1. Have a radiological and clinical diagnosis of OA based upon Arthritis Research Council (ACR) (Appendix 3) criteria affecting at least one knee of a minimum of 3 months in symptom duration prior to screening. An X-ray will be performed at screening if required.
   2. Have symptomatic OA of at least one knee. The symptoms should be significantly worse in one knee than the other if OA affects both knees.
   3. When questioned, confirm they experience moderate pain when climbing stairs.
   4. Be able to walk unaided or with the aid of one stick (2 sticks not allowed)
8. A minimum of 4 out 10 on the NRS (numerical rating scales) at screening and/ or a requirement for the use of an analgesic for the pain in the OA knee for most days during the previous three months. In addition, baseline pain must be stable for at least 72 hours prior to day 1 based on patient's assessment or day 1 may be delayed.
9. A maximum of 8 out of 10 on the NRS at screening. Enrollement may be delayed if, in the opinion of the investigator, the severity of pain represents an isolated incident.
10. In good general health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history or physical examination and suitable for treatment with both naproxen and paracetamol.

Exclusion Criteria:

* General

  1. The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines. However, a positive drug screen will not automatically exclude a subject if there is a valid explanation for the positive result other than drug abuse e.g. poppy seeds.
  2. History of regular alcohol consumption within 6 months of the study defined as:

     • An average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine.
  3. Intolerance of paracetamol or not response to Non Steriodal Anti Inflammatory Drugs (NSAID) therapy.
  4. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
  5. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
  6. Use of anticoagulants (warfarin, heparin) or anti-platelet aggregation agents (excluding low-dose aspirin) or a condition associated with decreased haemostasis.
  7. Use of prescription or non-prescription drugs within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety. Please also see OA exclusion criteria 10.
  8. Subject with a known allergy to or judged by the investigator not to be a suitable candidate for naproxen or paracetamol therapy based on medical history, concomitant medications, and concurrent systemic disease as described in the product labelling
  9. History or presence of gastro-intestinal, hepatic or renal disease or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs. In particular dyspepsia, peptic ulceration, gastrointestinal bleeding, ulcerative colitis or Crohn´s disease
  10. Presence of anaemia.
  11. Subjects who have asthma, have received anti-asthmatic medication within the last 5 years, have a history of NSAID-sensitive asthma or who have ever required hospital admission due to asthma.
  12. Presence of cardiac heart failure NYHA > 1.
  13. Presence of hypertension (BP systolic > 150 mmHg, diastolic > 90 mmHg) not adequately controlled by antihypertensive treatment.
  14. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
  15. Unwillingness or inability to follow the procedures outlined in the protocol including being able to undertake the walking as defined in the protocol.
  16. Inability or unwillingness to comply with study restrictions.

Exclusion criteria related to OA

1. Secondary causes of arthritis of the knee including septic arthritis, inflammatory joint disease, articular fracture, major dysplasias or congenital abnormality, ochronosis, acromegaly, hemochromatosis, Wilson's disease, and primary osteochondromatosis.
2. Had lower extremity surgery (including arthroscopy) within 6 months prior to screening or scheduled for surgery of any kind during the study period
3. Significant prior injury to the index knee within 12 months prior to screening.
4. Disease of the spine or other lower extremity joints of sufficient degree to affect the index knee.
5. Any other musculoskeletal or arthritic condition that may affect the interpretation of clinical efficacy and/or safety data or otherwise contraindicates participation in this clinical study (i.e., currently symptomatic fractures or any concurrent rheumatic disease such as but not limited to fibromyalgia, rheumatoid arthritis, and Reiter's syndrome are excluded).
6. Corticosteroid use prior to baseline as follows:

   * Intra-articular injection of steroids to the index knee within the previous 3 months
   * Intra-articular steroid injections into any site other than the index knee within the previous 1 month
   * Intra-muscular corticosteroid injections within the previous 3 months
   * Oral corticosteroids within the previous 1 month
7. Received hyaluronan injections into index knee within the previous six months prior to baseline.
8. Initiation of or change to an established physiotherapy program within 2 weeks prior to baseline or during the study period. An established physiotherapy program may be continued throughout the study period if unchanged in frequency and intensity.
9. Recent start or change in dose regimen ( 3 months prior to baseline) of any OA specific therapies (i.e., nutraceutical products) including but not limited to chondroitin or keratin sulfate, s-adenosyl methionine (SAMe) and glucosamine preparations.
10. Use of opioid analgesics other than codeine containing preparations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-09; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the time to ascend and descend 11 stairs | Screening, Day 1, Days 8,10,15,17,22,24

SECONDARY OUTCOMES:
Pain intensity difference as measured on numerical rating scales (NRS) after ascending and descending 11 stairs. | Screening, Day 1,Days 8,10,15,17,22,24
Change from baseline in the time to walk 20, 40 and 100m. | Screening, Day 1, Days 8,10,15,17,22,24
Pain intensity difference as measured on a numerical rating scales (NRS) after: 100m walk | Screening, Day 1, Days 8,10,15,17,22,24
Pain intensity difference as measured on a numerical rating scales (NRS) after: resting | Screening,Day 1, Days 2 to 7, 9, 11 to 14, 16, 18 to 21, 23, Days 8,10,15,17,22,24
Change from baseline in WOMAC scores | Day 1, Days 8,10,15,17,22,24
Patient Global Impression of Change (PGIC). | Days 8,10,15,17,22,24

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United Kingdom (3):
  - GSK Investigational Site, Buckshaw Village, Chorley, Lancashire
  - GSK Investigational Site, Cardiff
  - GSK Investigational Site, Manchester